CLINICAL TRIAL: NCT06409442
Title: Effects of Corrective External Support and Regional Vibration Applications Added to the Rehabilitation Program in Subacromial Pain Syndrome: Randomized Controlled Study
Brief Title: Effects of Corrective External Support and Regional Vibration Applications in Subacromial Pain Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Sevgi Sevi Yeşilyaprak, PhD, PT, Assoc. Prof., Dokuz Eylul University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 6920-GOA
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Subacromial Pain Syndrome
Keywords: shoulder impingement syndrome; pain; physical therapy and rehabilitation; ultrasonography
MeSH Terms: conditions — Shoulder Impingement Syndrome; Pain

STUDY DESIGN:
Intervention Model Description: Kinesio taping group (KTG), Local vibration therapy group (LVTG), and Control group (CG)
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (CG) (Standard Physiotherapy Program) (Active Comparator): Patients with subacromial pain syndrome will receive a 6-week treatment program. Patients will be given a treatment program by a physiotherapist three times a week, and on the other days, patients will practice six selected simple exercises at home.
  Standard Physiotherapy Program:
  The physiotherapy program will be given to all groups in the same way; It consists of patient education, Transcutaneous Electrical Nerve Stimulation (TENS) (20 minutes in each session), cold or hot pack application (15 minutes), mobilization and exercise program.
  Mobilization application is as follows:
  * Glenohumeral joint posterior glide
  * Glenohumeral joint inferior glide
  * Acromioclavicular joint inferior glide
  * Scapular mobilization
  The exercise program is as follows:
  * Phase 1 exercises
  * Phase 2 exercises
  * Phase 3 exercises
  Interventions: Other: Standard Physiotherapy Program
- Kinesio Taping Group (KTG) (Standard Physiotherapy Program + Kinesio Taping) (Active Comparator): In the group where kinesio taping will be added to Standard Physiotherapy Program, tape (Kinesio Tex, Standard 5 cm, KT-X-050, Tokyo, Japan) application will be performed by a certified physiotherapist. It will be used for 3 days, and the application will be repeated by the physiotherapist, the next day. Before taping, an allergic reaction test to the tape will be performed, if no allergy will be observed, participants will be taped and the tape maintenance brochure will be giving.
  Muscles for inhibition techniques:
  * Supraspinatus Muscle
  * Deltoid Muscle
  * Upper Trapezium Muscle
  Muscles for facilitation techniques:
  * Serratus Anterior Muscle
  * Lower Trapezium Muscle
  Interventions: Other: Standard Physiotherapy Program; Other: Kinesio Taping
- Local Vibration Therapy Group (LVTG) (Standard Physiotherapy Program + Local Vibration Therapy) (Experimental): In the LVT group, LVT via the Hypervolt™ (HYPERICE Inc, US) vibrating massage device will be added to Standard Physiotherapy Program. This device gives vibration with five different speed settings, vibrating at 3,200 percussions per minute. There are five different head options. The ball head attachment was chosen as it is the least aggressive option and the vibration from the device will be applied to the relevant muscle body. For the facilitator effect, high frequency application will be made to the lower trapezius and serratus anterior muscles. For the inhibitory effect, the upper trapezius, deltoid, pectoralis minor, and supraspinatus muscles will be applied at low frequency. The application will be 5 minutes for each muscle, for a total of 30 minutes. During the application, the speed will be controlled with a metronome, the travel time along the body of the relevant muscle will be 10 seconds, and the return time to the starting point will be 10 seconds.
  Interventions: Other: Standard Physiotherapy Program; Other: Local Vibration Therapy

INTERVENTIONS:
Other: Standard Physiotherapy Program — Patients with Subacromial Impingement Syndrome (SIS) will receive a 6-week treatment program. Patients will be given a physiotherapy treatment program by a physiotherapist three times a week, and on the other days, patients will practice six selected simple exercises at home.
Other: Kinesio Taping — In addition to the standard physiotherapy program, kinesio taping (device) will be applied.
  Arms: Kinesio Taping Group (KTG) (Standard Physiotherapy Program + Kinesio Taping)
Other: Local Vibration Therapy — In addition to the standard physiotherapy program, local vibration (device) will be applied.
  Arms: Local Vibration Therapy Group (LVTG) (Standard Physiotherapy Program + Local Vibration Therapy)

SUMMARY:
Sixty three individuals with chronic subacromial pain syndrome will be included in our study. In the evaluations to be made to the participants; Pain intensity will be measured with the Visual Analogue Scale (VAS), joint movement and shoulder proprioception will be measured with the inclinometer, and shoulder muscle strength will be measured with the digital hand dynamometer. In addition, functionality and disability levels will be determined by SPADI and Short form-Questionnaire for Arm, Shoulder and Hand Problems (Q-DASH). Supraspinatus tendon thickness and acromiohumeral space measurements will be made by ultrasonographic imaging. Patient satisfaction will be evaluated with the Visual Analog Patient Satisfaction Scale survey and quality of life will be evaluated with the SF-12 survey (The 12-item Short Form Survey).

Participants will be randomly divided into 3 groups of 21 participants each. In addition to the standard physiotherapy program, taping around the shoulder will be applied to the kinesio taping group, and localized vibration therapy around the shoulder will be applied to the localized vibration therapy group, in addition to the standard physiotherapy program. The Control Group (CG) will receive the same physiotherapy program as the other groups and will attend the same number of sessions as the other groups, accompanied by a physiotherapist. Evaluations will be made and analyzed before treatment, after 3 weeks of treatment, after 6 weeks of treatment, at 12 weeks and at the end of 24 weeks.

DETAILED DESCRIPTION:
The purpose of this study is to compare the effects of 6 week physiotherapy and kinesio taping (KT) combination (PKT) or physiotherapy and local vibration therapy (LVT) combination (PLVT) with physiotherapy program without these methods and with each other, after 3 weeks and 6 weeks of treatment, and to determine the differences in maintenance of their effects after 3 and 6 months. Shoulder pain is a common complaint that affects about one-third of individuals at some point in their lives. Subacromial Impingement Syndrome (SIS) is a non-infectious and often chronic disease that is the most common cause of shoulder pain. The incidence of the disease with age, its severity and the stage progress. Pain, loss of range of motion (ROM) and strength, functional limitations, and proprioceptive deficits are the findings of the disease. The changes in supraspinatus tendon thickness (SSTT) and narrowing in the subacromial space (SAS) are important parameters associated with these findings. SIS has a significant impact on the health-related quality of life (QoL) of patients, and the financial burden of the disease is high. Achieving and maintaining the treatment success for SIS is a challenging process due to the multi-factor pathogenesis and complexity of the joint. Exercise therapy is essential in treatment; however, some adjunct interventions could potentially improve treatment success. KT and LVT, which aim to optimize the muscle function and show similarities in terms of their facilitation and inhibition effects, have recently come to the fore in this context. Shoulder KT is used for reducing pain, improving function, proprioception, and SAS. However, there is moderate evidence that KT does not have beneficial effects over the sham-tape; studies have a high risk of bias, and acute or short-term results have been investigated with isolated applications. LVT is also used to improve muscle strength, ROM, and motor control. Portable and easy to use massage devices for LVT are on the agenda recently. However, in a single case report in the shoulder reported reduced pain, sensitivity, shoulder ROM, and increased muscle strength, but the results could not be generalized. It may be possible for LVT to improve pain, function, proprioception, and SAS, similar to KT. The positive effects of either method can positively affect the patients' satisfaction and QoL. Still, patient satisfaction has not been investigated before, and there is one investigation for the effects of KT on QoL. It is recommended to determine whether the addition of these methods to physiotherapy programs is more effective than the physiotherapy interventions without these methods with high-quality randomized controlled studies that have a high level of evidence (sufficient number of participants, sufficiently powered results, longer follow-up). Sixty three SIS patients will be included in this study. Short, medium, and long-term effects of 6 weeks PKT or PLVT will be compared objectively with each other and with a rehabilitation program without these methods. Shoulder pain will be evaluated with visual analog scale, ROM and proprioception with an inclinometer, muscle strength with the digital hand dynamometer, SSTT and SAS with ultrasonography, in addition, functionality and disability levels will be determined by SPADI and Short form-Questionnaire for Arm, Shoulder and Hand Problems (Q-DASH). And Patient satisfaction will be evaluated with the Visual Analog Patient Satisfaction Scale survey and quality of life will be evaluated with the SF-12 survey. The maintenance of the effects will be compared between the methods in long-term. Our study will be the first randomized controlled study having these characteristics. The investigators believe that it will contribute significantly to the literature, will help to choose the best management for SIS, the problematic treatment process will succeed in a shorter time and positive results last longer, useful information will be provided to the researchers and healthcare professionals for implementing rational treatment, therefore the success of SIS treatment can be increased, and it can contribute to the reduction of financial burdens.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study,
* Being over 18 years of age,
* Having diagnosed with subacromial impingement syndrome,
* SIS-related complaints have persisted for at least 3 months,
* Not having received any treatment for shoulder problems in the last 6 months,
* No history of shoulder injury other than subacromial impingement and/or shoulder symptoms requiring treatment for the last 1 year,
* To be able to read and write Turkish in order to complete all evaluations and applications in the study and to carry out evaluations that require reading and writing.

Exclusion Criteria:

* Having a history of fractures and surgery in the upper extremity and cervicothoracic region,
* Having another neurological, orthopedic or rheumatic shoulder problem such as frozen shoulder or instability,
* Having a systemic musculoskeletal disease,
* Known chest deformity, scoliosis diagnosis and physical disability,
* Presence of a skin problem or a condition that may be a contraindication to the application in the area where KT or LVT will be applied.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Shoulder Pain | Baseline, after 3 and 6 weeks of interventions period and then follow up measurement 3. and 6. months
  The level of pain felt during rest and activity will be marked on a 10 cm scale and the result will be recorded by measuring with a ruler. The value '0' means no pain; '10' indicates unbearable pain.
Range of Motion (Active and Pain-Free) | Baseline, and after 6 weeks of interventions period
  Active shoulder abduction, flexion, internal and external rotation movements will be measured using a 1-degree interval water-controlled inclinometer (Fabrication End Inc, NewYork, USA) while the patient is in the supine position.
  Pain-free joint range is the angle at which the patient first feels pain during active movement. Pain-free joint motion will be assessed by measuring pain-free joint motion during active shoulder elevation in the scapular plane with an inclinometer. While the patient is sitting in a chair with back support and lifts his arm up with his thumb pointing up, the angle at which he first feels pain will be recorded one degree below.
Muscle Strength | Baseline, and after 6 weeks of interventions period
  Change of trapezius,serratus anterior, supraspinatus and shoulder internal rotation isometric strength (in kg, with hand held dynamometer).The average of three consecutive repetitions will be recorded.
Shoulder Pain and Disability Index (SPADI) | Baseline, after 3 and 6 weeks of interventions period and then follow up measurement 3. and 6. months
  Shoulder Pain and Disability Index has 3 subscales: total, pain and disability. The pain subscale consists of 5 questions about shoulder pain during daily living activities, and the disability subscale consists of 8 questions about difficulty in performing daily living activities. A high score indicates increased pain and impaired shoulder function.To answer the questions, patients place a mark on a 10cm visual analogue scale for each question.The means of the two subscales are averaged to produce a total score ranging from 0 (best) to 100 (worst).
Short form-Questionnaire for Arm, Shoulder and Hand Problems (Q-DASH) | Baseline, after 3 and 6 weeks of interventions period and then follow up measurement 3. and 6. months
  The level of disability of the patients resulting from the upper extremity was determined by evaluating 11 different daily living activities. Each activity is scored between "1 = no difficulty" and "5 = not able to do it at all". In order for this score to be calculated, at least 10 out of 11 questions must be answered. Depending on the answers to the questions, a result score ranging from 0 (no disability)(best) to 100 (very serious disability)(worst) is calculated.
Quality of Life Assessment | Baseline, after 3 and 6 weeks of interventions period and then follow up measurement 3. and 6. months
  Short form 12-SF-12 survey will be used to evaluate quality of life. It assesses physical and mental health, the two main components of overall health. SF-12 consists of twelve questions. Mental and physical component scores will be calculated in accordance with the algorithm described by Ware.Scores can range from 16 to 112. A higher score indicates higher quality of life.

SECONDARY OUTCOMES:
Patient Satisfaction Rating | Baseline, after 3 and 6 weeks of interventions period and then follow up measurement 3. and 6. months
  The patient's symptom status (degree of improvement), physiotherapist (care provided) and overall satisfaction with the treatment will be evaluated by giving a score out of 10 with the Visual Analog Patient Satisfaction Scale. The lowest level individual is not satisfied at all; The highest level indicates that they are completely satisfied. In follow-up evaluations, only symptoms (degree of improvement) will be questioned.
Assessment of the Patient's Perceived Change in Condition | Baseline, after 3 and 6 weeks of interventions period and then follow up measurement 3. and 6. months
  The patient's perceived change in condition will be measured using the Global Change Rating Scale. This rating scale measures the person's perception of the change in their condition after treatment. The patient evaluates the overall change from the day he started treatment to the day he finished treatment using a 7-point Likert Scale. On the scale, a score of -7 would be scored as much, much worse, a score of 0 would be scored as almost the same, and a score of +7 would be scored as much, much better.
Ultrasonographic Measurements | Baseline, and after 6 weeks of interventions period
  Ultrasonographic measurements will be performed by examining images obtained in 2D using the LOGIQ e ultrasonography unit (LOGIQ e Ultrasound, GE(General Electric Company ) Healthcare, USA). A 7-12 megahertz(MHz) linear transducer will be used in the evaluations.
  To measure supraspinatus tendon thickness, the transducer will be placed perpendicular to the supraspinatus tendon in the anterior of the shoulder and two measurements will be made and the average will be taken. For acromiohumeral distance measurement, images of the humerus and acromion will be taken together at 0◦ and 60◦ scapular plane shoulder elevation, with the location of the transducer as the standard, 2.1 cm behind the first acromial arch in the coronal plane. It gives the shortest distance determined by 2D linear measurement between the acromion and humerus on the recorded images. The average of the measurements taken from the 1st and 2nd measurement locations will be recorded.
Proprioception | Baseline, and after 6 weeks of interventions period
  Change of shoulder abduction joint position sense (with digital inclinometer in degree) (Target angel:100 degree abduction). The target angle to be tested will be taught by the investigators with eyes open 3 times and eyes closed 3 times. The participant will then be asked to bring it to the target angle with their eyes closed. The deviation value from the target angle will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Sevgi Sevi Yeşilyaprak, PhD, Study Director — Dokuz Eylul University; Ezgi İrem Küçük, MSc Student, Study Chair — Dokuz Eylul University; Zana Gündüz, Bachelor's, Study Chair — Dokuz Eylul University; Mehmet Erduran, M.D, Study Chair — Dokuz Eylul University; Damla Karabay, PhD, Study Chair — İzmir Katip Çelebi University; Nursen İlçin, PhD, Study Chair — Dokuz Eylul University; Halime Ezgi Türksan, PhD Student, Study Chair — Dokuz Eylul University; Fatma Özden, PhD Student, Study Chair — Dokuz Eylul University
Locations (1):
- Dokuz Eylül University, Izmir, Balçova, Turkey (Türkiye)